CLINICAL TRIAL: NCT06612814
Title: PARP Inhibitor in Combination With CDK4/6 Inhibitor and Endocrine Therapy as the First-line Therapy for HR+/ HER2-Advanced Breast Cancer
Brief Title: PARP Inhibitor With CDK4/ 6 Inhibitor and Endocrine Therapy in HR+/ HER2-Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhimin Shao (Other)
Collaborators: First Hospital of China Medical University (Other); Sun Yat-sen University (Other); Chongqing University Cancer Hospital (Other); Fujian Medical University Union Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Shanghai First Maternity and Infant Hospital (Other); Affiliated Hospital of Nantong University (Other); Peking University Cancer Hospital & Institute (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Liaoning Cancer Hospital & Institute (Other); Northern Jiangsu People's Hospital (Other); Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhimin Shao, director, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N080
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — fluzoparib; dalpiciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): In this cohort, a patient would receive Dalpiciclib(CDK4/6 inhibitor) combined with Fluzoparib(Parp inhibitor) and endocrine therapy.
  Interventions: Drug: Fluzoparib; Drug: Dalpiciclib; Drug: Fulvestrant/AI
- Cohort 2 (Active Comparator): In this cohort, a patient would receive Dalpiciclib(CDK4/6 inhibitor) combined with endocrine therapy.
  Interventions: Drug: Dalpiciclib; Drug: Fulvestrant/AI

INTERVENTIONS:
Drug: Fluzoparib — Parp inhibitor
  Arms: Cohort 1
Drug: Dalpiciclib — CDK4/6 inhibitor
Drug: Fulvestrant/AI — Endocrine therapy

SUMMARY:
This study is a prospective, open-label, phase III clinical study for patients with HR+/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
Patients with SNF3 subtype of HR+/HER2- advanced breast cancer confirmed by the Department of Pathology and Key Laboratory of Breast Cancer of Fudan University Affiliated Cancer Hospital are planned to be enrolled. The main purpose is to evaluate the efficacy of PARP inhibitor in SNF3 subtype of HR+/HER2- advanced breast cancer in randomized controlled phase III clinical studies with larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥18 years and ≤ 75 years old;
* Histologically confirmed HR + / HER2- invasive breast cancer (specific definition: immunohistochemical detection of ER > 10% tumor cell positive is defined as ER positive, PR > 10% tumor cell positive is defined as PR positive, ER and / or PR Positive is defined as HR positive; HER2 0-1 + or HER2 is ++ but negative followed by FISH detection, no amplification, defined as HER2 negative);
* Subtype of similarity network fusion-3 (SNF-3) confirmed by the Department of Pathology and Key Laboratory of Breast Cancer of Fudan University Affiliated Cancer Hospital • Locally advanced breast cancer (incapable of radical local treatment) or recurrent metastatic breast cancer;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1); or unmeasurable lytic or mixed (osteolytic + osteoblastic) bone lesions in the absence of measurable lesions;
* Has adequate bone marrow function: absolute neutrophil count > 1.5x10ˆ9 /L; platelet count > 75x10ˆ9 /L, hemoglobin > 9g/dL;
* Patients had received no previous chemotherapy or targeted therapy for metastatic disease
* Has adequate liver function and kidney function: serum creatinine
* ECOG score ≤ 2 and life expectancy ≥ 3 months;
* Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

* Treatment with chemotherapy, radiotherapy, immunotherapy or surgery (outpatient clinic surgery excluded) for metastatic disease
* Symptomatic, untreated, or actively progressing CNS metastases(glucocorticoids or mannitol needed to control symptoms);
* Significant cardiovascular disease(including congestive heart failure, angina pectoris, myocardial infarction or ventricular arrhythmia in the last 6 months);
* is pregnant or breast feeding;
* Malignant tumors in the past five years (except cured skin basal cell carcinoma and cervical carcinoma in situ).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
ORR | andomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
CBR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5 years)
  the percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the participants.
OS | Randomization to death from any cause, through the end of study (approximately 5 years)
  time to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not provided